CLINICAL TRIAL: NCT07394127
Title: Effects of Inspiratory Muscle Training Combined With a Structured Swimming Program on Pulmonary Function and Asthma Control in Children With Mild Asthma: A Randomized Controlled Trial
Brief Title: Effects of Inspiratory Muscle Training Added to a Swimming Program in Children With Asthma
Acronym: IMT-SWIM-ASTHM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Coşkun YILMAZ, Director, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025/024
Record Dates: First submitted 2026-02-02; First posted 2026-02-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Asthma Control; Asthma; Asthma Chronic
Keywords: asthma control; pulmonary function; swimming; inspiratory muscle training; children; asthma
MeSH Terms: conditions — Asthma | interventions — Control Groups; Swimming

STUDY DESIGN:
Intervention Model Description: Intervention Model Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swimming Training Only (Control Group) (Other): Participants completed a supervised swimming training program for 4 weeks, consisting of three 60-minute sessions per week. Sessions included warm-up, main swimming exercises, and cool-down breathing exercises. Exercise intensity was maintained at approximately 65% of maximal heart rate.
  Interventions: Other: Swimming Training Only (Control Group); Other: Swimming + Inspiratory Muscle Training (Experimental Group)
- Swimming + Inspiratory Muscle Training (Experimental Group) (Experimental): Participants completed the same swimming training program as the control group. In addition, inspiratory muscle training was performed using a threshold pressure-loading device. IMT was conducted twice daily, starting at 30% of maximal inspiratory pressure and progressively increased by 5% weekly, over a 4-week period.
  Interventions: Other: Swimming Training Only (Control Group); Other: Swimming + Inspiratory Muscle Training (Experimental Group)

INTERVENTIONS:
Other: Swimming Training Only (Control Group) — Participants completed a supervised swimming training program for 4 weeks, consisting of three 60-minute sessions per week. Sessions included warm-up, main swimming exercises, and cool-down breathing exercises. Exercise intensity was maintained at approximately 65% of maximal heart rate.
Other: Swimming + Inspiratory Muscle Training (Experimental Group) — Participants completed the same swimming training program as the control group. In addition, inspiratory muscle training was performed using a threshold pressure-loading device. IMT was conducted twice daily, starting at 30% of maximal inspiratory pressure and progressively increased by 5% weekly, over a 4-week period.

SUMMARY:
This randomized controlled trial investigated the effects of adding inspiratory muscle training (IMT) to a structured swimming program on pulmonary function, respiratory muscle strength, ventilatory capacity, perceived exertion, and asthma control in children with mild persistent asthma. Thirty children aged 8-11 years were randomly assigned to either a swimming plus IMT group or a swimming-only group. Both groups participated in a supervised 4-week swimming program, while the experimental group additionally performed IMT twice daily. Pulmonary function tests, respiratory muscle strength, and Childhood Asthma Control Test (C-ACT) scores were assessed before and after the intervention.

DETAILED DESCRIPTION:
Asthma-related airway obstruction and respiratory muscle dysfunction may limit exercise tolerance and disease control in children. Swimming is considered a safe and beneficial exercise modality for pediatric asthma due to its humid environment and controlled breathing patterns. Inspiratory muscle training specifically targets respiratory muscle weakness and may further enhance pulmonary adaptations. This parallel-group randomized controlled trial examined whether combining IMT with swimming training yields superior improvements in lung function, respiratory muscle strength, ventilatory capacity, perceived exertion, and asthma control compared with swimming training alone. The intervention lasted four weeks, with objective pulmonary and respiratory muscle assessments conducted pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-11 years
* Clinically diagnosed mild persistent asthma according to GINA guidelines
* Baseline FEV₁ ≥ 80% predicted
* Stable asthma treatment for at least 4 weeks
* Written informed consent from parents or guardians

Exclusion Criteria:

* Mild intermittent, moderate, or severe persistent asthma
* Acute asthma exacerbation during the study
* Other chronic respiratory, cardiovascular, or neuromuscular diseases
* Recent upper respiratory tract infection
* Use of medications affecting pulmonary function other than standard asthma therapy

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure (MIP) | 4 weeks
  Measured using a handheld respiratory pressure device to assess inspiratory muscle strength.
Forced Expiratory Volume in 1 Second (FEV₁) | 4 weeks
  Assessed via spirometry to evaluate pulmonary function. Forced expiratory volume in one second (FEV₁) was measured using the spirometry method to assess lung function. FEV₁ values were reported as a percentage of the predicted value (% predicted) based on reference values. While there is no theoretical minimum or maximum limit for the measurement, higher FEV₁ values indicate better pulmonary function.
Childhood Asthma Control Test (C-ACT) Score | 4 weeks
  Validated questionnaire assessing asthma symptom control in children. The Childhood Asthma Control Test (C-ACT) is a self-report questionnaire used to assess the level of asthma symptom control in children over the past 4 weeks, with proven validity and reliability. The total scale score ranges from 0 to 27, with higher scores indicating better asthma control.

SECONDARY OUTCOMES:
Rating of Perceived Exertion (Borg Scale) | 4 week
  Rating of Perceived Exertion (Borg Scale), The Borg Rating of Perceived Exertion Scale (Borg Scale; 6-20) is a validated and reliable measure used to assess the level of exertion individuals perceive during exercise or physical activity over the past 4 weeks. Scale scores range from 6 to 20, with higher scores indicating a higher level of perceived exertion and, consequently, a poorer outcome.
Maximum Voluntary Ventilation (MVV) | 4 week
  Assessed via spirometry to evaluate pulmonary function. Maximum Voluntary Ventilation (MVV)
Peak Expiratory Flow (PEF) | 4 week
  Assessed via spirometry to evaluate pulmonary function. Peak Expiratory Flow (PEF)
Forced Vital Capacity (FVC) | 4 week
  Assessed via spirometry to evaluate pulmonary function. Forced Vital Capacity (FVC)

CONTACTS AND LOCATIONS:
Overall Officials: Coşkun YILMAZ, associate professor, Principal Investigator — Gümüşhane Universıty
Locations (1):
- Gumushane Univetsity, Gümüşhane, Trabzon, Ordu, Giresun, Rize, Artvin, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical restrictions and the inclusion of pediatric participants. Data sharing was not explicitly included in the informed consent, and sharing raw data could compromise participant confidentiality.